CLINICAL TRIAL: NCT01992055
Title: Functional Outcomes Following Neuropsychological Intervention in Acquired Brain Injury Outpatients With Executive Dysfunction
Brief Title: Outcomes Following Neuropsychological Intervention in Acquired Brain Injury Outpatients With Executive Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Lesley Ritchie, Assistant Professor/Neuropsychologist, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2013:389
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Acquired Brain Injury
Keywords: Executive dysfunction; Neuropsychological rehabilitation; Goal Management Training
MeSH Terms: conditions — Brain Injuries | interventions — Educational Status; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal Management Training (Experimental): The modified GMT intervention will consist of seven group sessions and, similar to van Hooren et al (2007), an individual session with a neuropsychologist on Session 5. Sessions will be held twice weekly. The manualized group sessions will include: (1) structured psychoeducation introducing participants to the brain and executive functioning, the relationship between stress and cognitive functioning, and relaxation training; (2) stepwise learning of GMT, including education regarding attentional lapses and goal neglect, as well as in-session practice targeting individual everyday functional deficits with the goal of maximizing generalization. Homework assignments targeting individual functional deficits will be assigned following each session.
  Interventions: Behavioral: Goal Management Training
- Education & relaxation training (Active Comparator): Education and relaxation training control group
  Interventions: Behavioral: Education & relaxation training

INTERVENTIONS:
Behavioral: Goal Management Training — Participants will be randomly assigned to the GMT Treatment. The GMT cognitive rehabilitation intervention program will be administered in group format, consisting of 8 sessions, including structured psychoeducation, relaxation training, and stepwise learning of GMT.
  Arms: Goal Management Training
Behavioral: Education & relaxation training — The Education & Relaxation Training Control Group program will also be administered in group format, consisting of two sessions, including structured psychoeducation and relaxation training. Participants assigned to the Control condition will be offered the opportunity to complete the full GMT program following the completion of the study.
  Arms: Education & relaxation training

SUMMARY:
This Clinical Trial is a pilot study being conducted to study the impact of a specific cognitive rehabilitation program, Goal Management Training (GMT), in adult patients with executive dysfunction and associated problems in everyday functioning. The intervention program will also include relaxation training and psychoeducation regarding brain injury on everyday functioning, emotional status, and executive functioning. Goal Management Training focuses on teaching individuals strategies to compensate for executive functioning deficits and is based on a theory of goal neglect resulting in disorganized behavior following frontal lobe injury. It emphasizes strategies for self-monitoring and self-evaluation in everyday life. Given its goal-oriented emphasis, focus on individual everyday difficulties, and reports of improvements in self-reported executive failures and mood, GMT appears to be an ideal intervention treatment for individuals with executive and functional deficits.

Given the emphasis of goal-oriented rehabilitation on reducing the impact of cognitive impairment on daily functioning, rather than attempting to restore cognitive abilities, a reduction in subjective reports of psychological distress is anticipated. This hypothesis is consistent with existing literature revealing reduced reports of annoyance and executive difficulties on self-report inventories. Improvements on tests of sustained attention and visuospatial problem-solving, as well as small effects on additional measures of planning, are also anticipated.

DETAILED DESCRIPTION:
Executive functions (EF) are higher-order cognitive processes used particularly under novel and complex conditions (Shallice, 1990) and comprise various abilities including devising goals, elucidating alternative solutions, implementing goal-directed behaviors, self-monitoring, and behavior modification and perseverance (Snyder, Nussbaum, & Robins, 2009). According to Sohlberg and Mateer (2001; p.234), EF may be described as cognitive abilities "required to complete goal-directed [behavior] that is not overlearned, automatic, and routine." As a result, executive dysfunction can impair one's ability to function independently (Bolognani et al., 2007). Research has identified a positive relationship between functional ability and EF (Hanks, Rapport, Millis, & Deshpande, 1999). Additionally, differential declines in EF are observed in normal aging after the age of 60 years (Treitz, Heyder, & Daum, 2007). As well, the profile of cognitive impairment in Parkinson's disease is marked by a predominance of executive dysfunction, followed by memory deficits (Emre, 2003; Emre, 2004; Verbaan et al, 2007). In addition to traumatic and acquired brain injuries, executive dysfunction and functional deficits have been observed in individuals with psychiatric illnesses such as ADHD (Attention Deficit Hyperactivity Disorder; e.g., Willcutt, Doyle, Nigg, Faraone, & Pennington, 2005), psychostimulant and opioid abuse (e.g., Verdejo-Garcıa, Lopez-Torrecillas, Aguilar de Arcos, & Perez-Garcıa, 2005; Fernández-Serranoa, Pérez-García, & Verdejo-García, 2011), bipolar disorder (e.g., Frangou, Donaldson, Hadjulis, Landay, & Goldstein, 2005; Maalouf et al., 2010), and geriatric depression (Lockwood, Alexopoulos, van Gorp, 2002). The prominence of executive dysfunction in individuals with acquired brain injury and mental illness, and the associated costs on the healthcare system, highlights a role for cognitive rehabilitation.

Cognitive rehabilitation refers to interventions aiming to enhance or support cognitive abilities following brain injury, with an emphasis on achieving functional changes. It is a structured, goal-oriented, collaborative process between the therapist and the patient (and, where possible, caregivers/family) and is informed by medical and neuropsychological data (Sohlberg & Mateer, 2001). A recent meta-analysis of the effectiveness of cognitive rehabilitation following acquired brain injury revealed a significant effect on global cognitive functioning, with time-since-injury acting as a moderating variable. Attention training following traumatic brain injury (TBI) and language and visuospatial training for aphasia were identified as effective treatments (Rohling, Faust, Beverly, & Damaskis, 2009). In their review of intervention approaches for executive dysfunction, Boelen, Spikman, and Fasotti (2011) describe three approaches used in previous studies. First, compensatory strategies emphasize teaching patients cognitive strategies to offset cognitive deficits. Second, restorative strategies aim to repair cognitive functions. Third, behavioral therapy interventions seek to modify behavior through means such as token economies.

An example of the compensatory approach to executive dysfunction is Goal Management Training (GMT). GMT is a cognitive rehabilitation strategy based on Duncan's (1986) theory of goal neglect resulting in disorganized behavior following frontal lobe injury. It emphasizes strategies for self-monitoring and self-evaluation in everyday life, including pausing, identifying the task at hand, outlining the goals and listing the required steps, completing the task, and evaluating the successful completion of the task.

Given the relationship between disorganized behavior and functional dependence, the use of GMT in patients with executive dysfunction is highly relevant. Levine et al. (2000) compared the effectiveness of GMT and motor skills training (MST) in patients with TBI who were living independently in the community. The GMT group exhibited improved performance on paper and pencil tasks (e.g., proofreading) and slowed speed of task completion suggested increased attention to task demands. Improvements on the MST trained tasks were noted for the MST group. Fish and colleagues (2007) evaluated the effect of a "content-free" cueing strategy (i.e., text messages reading STOP!), the first stage in GMT, to compensate for goal-neglect following brain injury. The authors reported significant improvements in goal-directed behavior with the addition of "content free" cues and conclude that the provision of cues improves goal management by increasing self-monitoring.

GMT has also been evaluated in normal aging, given the relationship between reduced executive functioning, functional difficulties, and aging. Van Hooren and colleagues (2007) evaluated 69 Dutch adults aged 55 years or older for the impact of a structured 12-session GMT program on cognitive functioning, self-reported mood, and self-reported cognitive complaints and failures. Their GMT program included psychoeducation regarding cognitive functioning and functional difficulties and their study design utilized a randomized wait-list control group. The results revealed reduced annoyance, improved management of cognitive failures, and decreased anxiety in the treatment group, relative to controls. No improvement on objective measures of cognitive functioning was noted. In another wait-list controlled study evaluating GMT in normal aging, Levine and colleagues (2007) reported decreased self-report of executive failures and improved performance on simulated real-life tasks in 49 healthy older adults.

In addition to group studies, GMT has been evaluated in single case studies. Schweizer et al (2008) provided seven, weekly, two-hour sessions of GMT to a patient with focal damage to the cerebellum. Evaluation of the treatment included pre-, post-, and long-term (i.e., 4 months post-intervention) administration of attention, executive functioning, and self-report measures. Although modest improvements on objective measures of executive functioning were observed, the patient endorsed significant improvements in functional abilities (i.e., return to work). Similarly, Levine and colleagues (2000) observed improvements in meal preparation, following two sessions of GMT, in a patient in the chronic stage of recovery from meningo-encephalitis. The GMT sessions focused on the five stages of GMT using the patient's recipes as training examples. The effect of GMT on meal preparation was maintained at a six-month follow-up evaluation.

Recently, the first controlled, partially randomized, study of GMT was completed with patients in the chronic stage of recovery from a focal brain injury and who were exhibiting persistent executive dysfunction (Levine et al., 2011). Significant improvements in sustained attention, behavioral consistency, and problem-solving were reported for the GMT group, with no significant effects found for the control group. However, in contrast to previous studies (Levine et al., 2007; van Hooren et al., 2007), no change on self-report measures of everyday executive functioning was observed. The authors attribute the lack of change in subjective report to two possible factors: 1) an absence of collateral ratings and 2) reduced insight due to executive dysfunction or improved insight resulting in increased item endorsement. The authors conclude that GMT is an effective intervention for executive dysfunction, which produces improvements in both trained and untrained behaviors.

Goal management training has been described as a unique cognitive rehabilitation technique, given its theoretical basis in goal neglect following frontal lobe damage and its emphasis on real-life behaviors (Levine et al., 2000). The authors also reveal that, for rehabilitation strategies to generalize to other behaviors, generalization must be a component of the intervention itself. This conclusion is consistent with Sohlberg and Mateer's (2001) suggestion that clinicians should "program generalization" by training overlearning and general strategies for various locations and tasks, emphasizing individual difficulties, incorporating significant others in the rehabilitation process, and planning for obstacles. It has been recommended that rehabilitation for executive dysfunction emphasize the achievement of independence in functional activities and generalization to everyday activities (Boelen, Spikman, & Fasotti, 2011). Given its goal-oriented emphasis, focus on individual everyday difficulties, and reports of improvements in self-reported executive failures and mood, GMT appears to be an ideal intervention for individuals with functional and executive function impairment.

OBJECTIVES

The purpose of the proposed study is to evaluate the effectiveness of a GMT group, emphasizing compensatory strategies for executive dysfunction (e.g., goal neglect and attentional lapses), as well as relaxation training and psychoeducation regarding brain injury, in a sample of adult outpatients with identified executive dysfunction and associated functional deficits. Specific objectives include:

1. Evaluation of the short-term efficacy of GMT on self- and collateral-report of everyday functioning.
2. Evaluation of the short-term efficacy of GMT on neuropsychological outcome measures.
3. Evaluation of the long-term (i.e., 1 year) efficacy of GMT on self- and collateral-report of everyday functioning.
4. Identification of neuropsychological measures sensitive to cognitive change following GMT, through the use of a more extensive battery of neuropsychological tests, compared to previous studies.
5. Evaluation of the long-term (i.e., 1 year) efficacy of GMT on neuropsychological outcome measures.
6. Identify the primary mediator of change in GMT by comparing a control group receiving two sessions of relaxation training and psychoeducation relative to a treatment group receiving the complete GMT program (including relaxation training and psychoeducation).

HYPOTHESES Given the emphasis of goal-oriented rehabilitation on reducing the impact of cognitive impairment on daily functioning, rather than attempting to restore cognitive abilities, a reduction in subjective reports of psychological distress is anticipated. This hypothesis is consistent with existing literature revealing reduced reports of annoyance and executive difficulties on self-report inventories (van Hooren et al., 2007; Levine et al., 2007). Previous research has identified improvement on sustained attention and visuospatial problem-solving tasks following GMT (Levine et al., 2011). The proposed battery of neuropsychological tests includes a greater number of neuropsychological measures evaluating different neuropsychological functions. Improvements on tests of sustained attention and visuospatial problem-solving, as well as small effects on additional measures of planning, are also anticipated.

METHODOLOGY Participants Group Assignment Participants will be randomly assigned to a GMT Treatment or Control Group. The GMT cognitive rehabilitation intervention program will be administered in group format, consisting of 8 sessions, including structured psychoeducation, relaxation training, and stepwise learning of GMT. The Control Group program will also be administered in group format, consisting of two sessions, including structured psychoeducation and relaxation training. Participants assigned to the Control condition will be offered the opportunity to complete the full GMT program following the completion of the study.

Intake: A screening interview with the patient and their significant other will be conducted to gather essential background demographic and medical information, including self- and collateral-report of cognitive, emotional, and functional status. Participants referred without a baseline neuropsychological assessment will undergo a standardized neuropsychological battery. For patients referred with a brief cognitive screen, additional neuropsychological measures will be administered.

GMT Treatment Group: A modified (i.e., including psychoeducation and relaxation training) GMT cognitive rehabilitation intervention program will be administered in group format. Each group will consist of six participants to ensure sufficient time to address both group and individual functional difficulties. Although more cost-effective, larger groups of patients with executive dysfunction are not planned, given the prominence of organizational and attention deficits among patients with executive dysfunction. The modified GMT intervention will consist of seven group sessions and, similar to van Hooren et al (2007), an individual session with a neuropsychologist on Session 5. Sessions will be held twice weekly. The manualized group sessions will include: (1) structured psychoeducation introducing participants to the brain and executive functioning, the relationship between stress and cognitive functioning, and relaxation training; (2) stepwise learning of GMT, including education regarding attentional lapses and goal neglect, as well as in-session practice targeting individual everyday functional deficits with the goal of maximizing generalization. Homework assignments targeting individual functional deficits will be assigned following each session.

Control Group: Participants randomly assigned to the Control condition will participate in two group sessions emphasizing psychoeducation and relaxation training. The proposed Control condition goes beyond the current standard of care, which does not include any cognitive or psychological intervention beyond neuropsychological and medical assessment. In keeping with the GMT Treatment group, the Control groups will consist of six participants. Sessions will be scheduled along side the GMT Treatment sessions (i.e., two sessions in one week)

ELIGIBILITY:
Inclusion Criteria:

* Participants may be included in the study if they are identified as having EF impairments, secondary to an acquired brain injury, and are between the ages of 18 and 65 years. Informed consent will be gathered from each participant. Eligible participants will be informed about the purpose of the study, the associated risks and benefits, and their option to withdraw from the study at any time without penalty. Potential risks include subtle discomfort when initially participating in relaxation exercises, which typically resolves with familiarity, and mild distress during neuropsychological assessment. These issues sometimes arise during standard clinical practice and the neuropsychologists involved are experienced in assisting people in reducing their distress.

Exclusion Criteria:

* Individuals with significant memory impairment, receptive language deficits, active psychosis, severe depression (i.e., Beck Depression Inventory - II [BDI-II] ≥ 30), or a diagnosis of dementia will be excluded from participating in the study.. A minimum of 36 participants will be recruited for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in neuropsychological functioning at 1 week post-intervention | 1 week post-intervention
  Change in test scores on the following measures:
  Connor's Continuous Performance Test - II Delis-Kaplan Executive Functioning Scale Tower Test Trail Making Test Ruff Figural Fluency Test Controlled Oral Word Association Test Semantic Fluency Golden's Stroop Color and Word Test BADS Six Elements Test Brief-A Self and Family Report Inventories SCL-90-R Self-Report Inventory Word Memory Test Medical Symptom Validity Test (MSVT) Non-Verbal MSVT

SECONDARY OUTCOMES:
Change from Baseline in neuropsychological functioning at 4 weeks post-intervention | 4 weeks post-intervention
  Change in test scores on the following measures:
  Connor's Continuous Performance Test - II Delis-Kaplan Executive Functioning Scale Tower Test Trail Making Test Ruff Figural Fluency Test Controlled Oral Word Association Test Semantic Fluency Golden's Stroop Color and Word Test BADS Six Elements Test Brief-A Self and Family Report Inventories SCL-90-R Self-Report Inventory Word Memory Test Medical Symptom Validity Test Non-Verbal MSVT

OTHER OUTCOMES:
Change from Baseline in neuropsychological functioning at 1 year post-intervention | 1 year post intervention
  Change in test scores on the following measures:
  Connor's Continuous Performance Test - II Delis-Kaplan Executive Functioning Scale Tower Test Trail Making Test Ruff Figural Fluency Test Controlled Oral Word Association Test Semantic Fluency Golden's Stroop Color and Word Test BADS Six Elements Test Brief-A Self and Family Report Inventories SCL-90-R Self-Report Inventory Word Memory Test Medical Symptom Validity Test Non-Verbal MSVT

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Ritchie, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada